Official Title Azacitidine (AZA) Combined With N-

Acetyl-L-cysteine (NAC) for Prolonged

Isolated Thrombocytopenia (PIT) After

Hematopoietic Stem Cell

Transplantation (HSCT)

**NCT Number** 

Date of the document 11/1/2021

## Informed Consent Form

Azacitidine (AZA) Combined With N-Acetyl-L-cysteine (NAC) for Prolonged Isolated Thrombocytopenia (PIT) After Hematopoietic Stem Cell Transplantation (HSCT)

#### Dear Madam/Sir,

You will be invited to participate in a clinical study. The following items describe the research background, purpose, methods, benefits, discomforts, inconveniences and your rights and interests of this study. Please read them carefully before you participate in the clinical study. This Informed Consent provides you with information to help you decide whether or not to participate in this clinical study. If you have any questions, please ask the physician in charge of the study to ensure that you fully understand the relevant information. Your participation in this study is voluntary. If you agree to participate in this clinical study, please sign on the signature page of the informed consent.

### 1. Background

Prolonged isolated thrombocytopenia (PIT) after allogeneic hematopoietic stem cell transplantation (HSCT) is one of the most common complications after transplantation, with an incidence of 5-44%, including primary thrombocytopenia and secondary thrombocytopenia. However,PIT often leads to fatal bleeding, increasing transplant-related mortality and seriously affecting the quality of life of patients.

So far, no standard treatments for PIT have been implemented. Commonly used treatments are ranging from glucocorticoid, human recombinant platelet hormone, human recombinant interleukin - 11, to intravenous immunoglobulin, but the above treatment response rate between patients demonstrates heterogeneity. Besides, once the treatment is invalid, it always results in poor prognosis. In order to prevent bleeding, platelet infusion is needed in most patients, but platelet infusion may also lead to many adverse reactions, such as acute lung injury, heart failure, viral infection, etc., and ineffective infusion may occur in some patients. Therefore, platelet infusion cannot be used as a means of long-term bleeding prevention. For patients diagnosed with PIT, there is an urgent need to find new therapies to improve the outcome.

Previous studies of our center revealed that in patients with poor platelet reconstruction after transplantation, the application of low-dose Decitabin (DAC) can effectively promote the reconstruction of megakaryocytes. Meanwhile, it was found that N-acetyl-L-cysteine (NAC) can improve the oxidative microenvironment of bone marrow and further promote the reconstruction of megakaryocytes. The transplantation data of our center in the past 2 years showed that the application of Azacytidine (AZA) after transplantation similarly promoted the implantation of megakaryocytes in patients with poor platelet reconstruction after transplantation, and the myelosuppression period was shorter.

# 2. Purpose of the study

This clinical trial is a multicenter, prospective, double-armed study. The main purpose of this clinical trial is to observe the efficacy and safety of Aza combined with NAC in the treatment

of PIT, and to provide evidence for the use of Aza combined with NAC in patients.

## 3. Mothods of the study

After you sign the Informed Consent Form, you will receive AZA combined with NAC treatment if you are eligible for inclusion after screening. The duration of the study will be 12 weeks, with AZA at 50mg day 1-5 subcutaneously and NAC at 600mg day 1-28 orally, in a 28-day cycle. The endpoint was assessed after 3 cycles of treatment. During the study period, you will need to be followed up once a week for blood tests. The specific follow-up time can comply with the clinician's arrangement.

# 4. Possible benefits for participating in the study

AZA in combination with NAC offers a new treatment option with the potential to promote platelet implantation in patients with PIT.

- 5. Possible risks and discomforts associated with participating in the study Common adverse reactions include bone marrow suppression, headache, bruising, infection, bleeding, fatigue, etc.
- 6. Treatment and financial compensation for study-related injuries
  If you have CTCAE grade III-IV adverse reactions during the study period, the study will be
  immediately stopped and you will receive appropriate rescue measures. If you are harmed
  in connection with the study, the researchers will bear the relevant medical expenses and
  corresponding economic compensation in accordance with the relevant laws and
  regulations of our country.

#### 7. Routine treatment options

The current treatment for PIT can be treated with human recombinant thrombopoietin (RHTPO), which in turn increases the risk of thrombosis in the user.

#### 8. Rights for participators

You shall have the following rights during the process of participating in the clinical trial, including voluntary participation and withdrawal at any time, as well as no discrimination or retaliation against you after withdrawal at any time and no impact on your medical treatments.

## 9. Confidentiality of your data

The Investigator is responsible for handling your research data in accordance with applicable data protection regulations. However, such information can be accessed by the Ethics Committee and higher administrative departments during inspections. The results may all be presented in medical journals/conferences, but your identity will not be disclosed.

By signing this Informed Consent Form, your health information will be used by the physician and the staff involved in this study. Your authorization will allow us to use your health information till the end of this study. However, you may withdraw the informed

consent form at any time through the study from the responsible physician.

My statement: I have read this informed consent carefully. My questions have been answered. I understand that participation in this study is voluntary, and I can choose not to participate in this study, or I can withdraw from the study after notifying the researcher at any time without discrimination or retaliation, and my medical treatment and rights and interests will not be affected by this.

If I require additional treatment, or I do not comply with the study plan, or for any other reasonable reason, the study physician may discontinue my participation of the study. I voluntarily agree to participate in the clinical study and I will receive a signed copy of the "Informed Consent Form".

| Please sign here | | |
|------------------|----|----|
| Date | /_ | /_ |